CLINICAL TRIAL: NCT03656939
Title: AN OBSERVATIONAL SAFETY STUDY FOR PREVENAR 13 AMONG CHINESE CHILDREN
Brief Title: A Safety Study For Prevenar 13 Among Chinese Children
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851193
Record Dates: First submitted 2018-07-20; First posted 2018-09-04 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: Seizures; Urticaria and Angioedema; Apnea; Fever
MeSH Terms: conditions — Seizures; Urticaria; Angioedema; Apnea; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prevenar 13 cohort: This is a non-interventional study. Children in the study receive Prevenar 13 per normal medical practice.

SUMMARY:
This is an observational study based on a population-based EHR database.

DETAILED DESCRIPTION:
This observational study based on a population-based EHR database in Yinzhou district of Ningbo city in China is to estimate incidence rates of seizures (including febrile seizures), urticaria and angioedema, apnea, and fever among Chinese children after receiving Prevenar 13. In addition, a validation study including validation of International classification of diseases, tenth revision (ICD-10) codes or ICD-10 code based algorithm for identifying all safety outcomes of interest and a prospective cohort study in a sub-population of the main study will be conducted in order to offset the potential biased results from the main study because of potential misclassification of the safety outcomes of interest due to miscoding and/or undercoding of ICD-10 codes used to identify these safety outcomes in the EHR database.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the main study, children in Yinzhou population-based EHR database must be aged 1 to 24 months and receive at least one dose of 13vPnC between May 1st, 2017 and July 24th, 2020 where the first dose is received before or on July 24th, 2020 since a 7-day post-vaccination follow-up for each dose in each child receiving 13vPnC is needed. For the prospective cohort in a sub-population of the main study, eligible children for the main study must receive the first dose of 13vPnC between August 1st, 2018 and July 24th, 2020 and an informed consent must be obtained from parents/legal guardians.

Exclusion Criteria:

There are no exclusion criteria for this study.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The main study population consists of eligible children aged 1-24 months receiving at least one dose of 13vPnC recorded in Yinzhou EHR database between May 1st, 2017 and July 24th, 2020 (ie, one week prior to the end of the study).
  For the prospective cohort in a sub-population of the main study, eligible children for the main study must receive the first dose of 13vPnC between August 1st, 2018 and July 24th, 2020. It should be noted that the actual start date for the prospective cohort study is pending on the approval of Human Genetic Resources Administration of China (HGRAC) application.
Sampling Method: Non-Probability Sample
Enrollment: 21240 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- School of Public Health at Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study had main study and prospective cohort study. Data for main study and prospective cohort study were observed during 2 years of this observational study.
Pre-assignment Details: The main study utilized population-based Yinzhou electronic health record (EHR) database. As part of validation study, prospective cohort study was conducted in sub-population of main study. Main study included eligible children aged 1-24 months who received at least 1 dose of Prevenar 13 recorded in Yinzhou EHR database between 1 May 2017 and 24 July 2020. Prospective cohort study had eligible children for main study who received first dose of Prevenar 13 between 1 August 2018 and 24 July 2020.
Groups:
- Prevenar 13: Main study cohort included participants aged 1 to 24 months who received at least 1 dose of Prevenar 13 between 1 May 2017 and 24 July 2020 in the Yinzhou database were observed in the study. First dose of Prevenar 13 was received on or before 24 July 2020. Prospective study cohort included eligible participants of the main study who received first dose of Prevenar 13 between 1 August 2018 and 24 July 2020 in the Yinzhou EHR database were observed. Participants were followed up to 7 days after each dose of Prevenar 13.
Period: Overall Study
Arm/Group | Prevenar 13
Started | 21240
Main Study Cohort | 21240
Main Study Cohort: Participants Who Received Dose 1 | 20318
Main Study Cohort: Participants Who Received Dose 2 | 19387
Main Study Cohort: Participants Who Received Dose 3 | 18415
Main Study Cohort: Participants Who Received Dose 4 | 12944
Prospective Study Cohort | 2300
Prospective Study Cohort: Participants Who Received Dose 1 | 2300
Prospective Study Cohort: Participants Who Received Dose 2 | 2203
Prospective Study Cohort: Participants Who Received Dose 3 | 2047
Prospective Study Cohort: Participants Who Received Dose 4 | 1291
Completed | 21240
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the main study population which consisted of eligible children aged 1-24 months who received at least 1 dose of Prevenar 13 recorded in Yinzhou EHR database between 1 May 2017 and 24 July 2020.
Arm/Group | Prevenar 13
Number analyzed (Participants) | 21240
Age, Continuous [Mean (Standard Deviation); unit: Months] | 3.15 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9944
  Male | 11296
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of all seizures events experienced during the specified risk window (0-3 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Groups:
- Prevenar 13: Main Study Cohort: Participants aged 1 to 24 months who received at least 1 dose of Prevenar 13 between 1 May 2017 and 24 July 2020 in the Yinzhou database were observed in the study. First dose of Prevenar 13 was received on or before 24 July 2020. Participants were followed up to 7 days after each dose of Prevenar 13.
- Prevenar 13 Cohort: Prospective Cohort Study: In this cohort, eligible participants of the main study who received first dose of Prevenar 13 between 1 August 2018 and 24 July 2020 in the Yinzhou EHR database were observed. Participants were followed up to 7 days after each dose of Prevenar 13.
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81272 | 9200
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

2. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of all seizures events experienced during the specified risk window (4-7 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81269 | 9200
Events per 1000 person-days | 0.025 [0.006 to 0.098] | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

3. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of all seizures events experienced during the specified risk window (0-7 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 162541 | 18400
Events per 1000 person-days | 0.012 [0.003 to 0.049] | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

4. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of febrile seizures events experienced during the specified risk window (0-3 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81272 | 9200
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

5. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of febrile seizures events experienced during the specified risk window (4-7 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81271 | 9200
Events per 1000 person-days | 0.012 [0.002 to 0.087] | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

6. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of febrile seizures events experienced during the specified risk window (0-7 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 162543 | 18400
Events per 1000 person-days | 0.006 [0.001 to 0.044] | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

7. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of urticaria and angioedema events experienced during the specified risk window (0-3 days post-vaccination) divided by the observed time at risk, multiply by 1000. Urticaria represents an allergic reaction. Angioedema is an area of swelling (edema) of the lower layer of skin and tissue just under the skin or mucous membranes.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81269 | 9197
Events per 1000 person-days
  Urticaria | 0.012 [0.002 to 0.087] | 0.326 [0.105 to 1.011]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

8. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of urticaria and angioedema events experienced during the specified risk window (4-7 days post-vaccination) divided by the observed time at risk, multiply by 1000. Urticaria represents an allergic reaction. Angioedema is an area of swelling (edema) of the lower layer of skin and tissue just under the skin or mucous membranes.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81267 | 9200
Events per 1000 person-days
  Urticaria | 0.025 [0.006 to 0.098] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

9. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of urticaria and angioedema events experienced during the specified risk window (0-7 days post-vaccination) divided by the observed time at risk, multiply by 1000. Urticaria represents an allergic reaction. Angioedema is an area of swelling (edema) of the lower layer of skin and tissue just under the skin or mucous membranes.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 162532 | 18385
Events per 1000 person-days
  Urticaria | 0.019 [0.006 to 0.057] | 0.163 [0.053 to 0.506]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

10. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of apnea events experienced during the specified risk window (0-3 days post-vaccination) divided by the observed time at risk, multiply by 1000. Apnea is the cessation of breathing.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81272 | 9200
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

11. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of apnea events experienced during the specified risk window (4-7 days post-vaccination) divided by the observed time at risk, multiply by 1000. Apnea is the cessation of breathing.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81272 | 9200
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

12. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of apnea events experienced during the specified risk window (0-7 days post-vaccination) divided by the observed time at risk, multiply by 1000. Apnea is the cessation of breathing.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 162544 | 18400
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

13. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of fever events experienced during the specified risk window (0-3 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81137 | 8888
Events per 1000 person-days | 0.555 [0.414 to 0.743] | 10.689 [8.742 to 13.07]

14. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of fever events experienced during the specified risk window (4-7 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 81265 | 9195
Events per 1000 person-days | 0.049 [0.019 to 0.131] | 0.544 [0.226 to 1.307]

15. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of fever events experienced during the specified risk window (0-7 days post-vaccination) divided by the observed time at risk, multiply by 1000.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 162223 | 17702
Events per 1000 person-days | 0.296 [0.223 to 0.393] | 5.649 [4.644 to 6.872]

16. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 3 Days After Dose 2
Description: as for outcome 1
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77548 | 8812
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

17. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 4 to 7 Days After Dose 2
Description: as for outcome 2
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77548 | 8812
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

18. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 7 Days After Dose 2
Description: as for outcome 3
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 155096 | 17624
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

19. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 3 Days After Dose 2
Description: as for outcome 4
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77548 | 8812
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

20. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 4 to 7 Days After Dose 2
Description: as for outcome 5
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77548 | 8812
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

21. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 7 Days After Dose 2
Description: as for outcome 6
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 155096 | 17624
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

22. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 3 Days After Dose 2
Description: as for outcome 7
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77536 | 8808
Events per 1000 person-days
  Urticaria | 0.065 [0.027 to 0.155] | 0.227 [0.057 to 0.908]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

23. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 4 to 7 Days After Dose 2
Description: as for outcome 8
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77530 | 8812
Events per 1000 person-days
  Urticaria | 0.129 [0.069 to 0.240] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

24. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 7 Days After Dose 2
Description: as for outcome 9
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 155046 | 17612
Events per 1000 person-days
  Urticaria | 0.097 [0.058 to 0.161] | 0.114 [0.028 to 0.454]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

25. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 3 Days After Dose 2
Description: as for outcome 10
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77548 | 8812
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

26. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 4 to 7 Days After Dose 2
Description: as for outcome 11
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77548 | 8812
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

27. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 7 Days After Dose 2
Description: as for outcome 12
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 155096 | 17624
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

28. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 3 Days After Dose 2
Description: as for outcome 13
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77439 | 8696
Events per 1000 person-days | 0.517 [0.379 to 0.704] | 4.14 [2.986 to 5.739]

29. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 4 to 7 Days After Dose 2
Description: as for outcome 14
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 77531 | 8808
Events per 1000 person-days | 0.116 [0.060 to 0.223] | 0.568 [0.236 to 1.364]

30. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 7 Days After Dose 2
Description: as for outcome 15
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Person days at risk) | 154811 | 17360
Events per 1000 person-days | 0.310 [0.234 to 0.411] | 2.362 [1.739 to 3.208]

31. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 3 Days After Dose 3
Description: as for outcome 1
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73660 | 8188
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

32. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 4 to 7 Days After Dose 3
Description: as for outcome 2
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73660 | 8188
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

33. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 7 Days After Dose 3
Description: as for outcome 3
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 147320 | 16376
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

34. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 3 Days After Dose 3
Description: as for outcome 4
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73660 | 8188
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

35. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 4 to 7 Days After Dose 3
Description: as for outcome 5
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73660 | 8188
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

36. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 7 Days After Dose 3
Description: as for outcome 6
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 147320 | 16376
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

37. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 3 Days After Dose 3
Description: as for outcome 7
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73657 | 8188
Events per 1000 person-days
  Urticaria | 0.054 [0.020 to 0.145] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

38. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 4 to 7 Days After Dose 3
Description: as for outcome 8
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73638 | 8188
Events per 1000 person-days
  Urticaria | 0.136 [0.073 to 0.252] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

39. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 7 Days After Dose 3
Description: as for outcome 9
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 147279 | 16376
Events per 1000 person-days
  Urticaria | 0.095 [0.056 to 0.161] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

40. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 3 Days After Dose 3
Description: as for outcome 10
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73660 | 8188
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

41. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 4 to 7 Days After Dose 3
Description: as for outcome 11
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73660 | 8188
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

42. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 7 Days After Dose 3
Description: as for outcome 12
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 147320 | 16376
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

43. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 3 Days After Dose 3
Description: as for outcome 13
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73601 | 8115
Events per 1000 person-days | 0.367 [0.252 to 0.535] | 2.834 [1.884 to 4.265]

44. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 4 to 7 Days After Dose 3
Description: as for outcome 14
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 73634 | 8180
Events per 1000 person-days | 0.190 [0.113 to 0.321] | 0.489 [0.184 to 1.303]

45. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 7 Days After Dose 3
Description: as for outcome 15
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Person days at risk) | 147127 | 16206
Events per 1000 person-days | 0.279 [0.205 to 0.379] | 1.604 [1.092 to 2.356]

46. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 3 Days After Dose 4
Description: as for outcome 1
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51766 | 5164
Events per 1000 person-days | 0.058 [0.019 to 0.180] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

47. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 4 to 7 Days After Dose 4
Description: as for outcome 2
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51775 | 5164
Events per 1000 person-days | 0.039 [0.010 to 0.155] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

48. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 7 Days After Dose 4
Description: as for outcome 3
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 103529 | 10328
Events per 1000 person-days | 0.048 [0.020 to 0.116] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

49. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 3 Days After Dose 4
Description: as for outcome 4
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51776 | 5164
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

50. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 4 to 7 Days After Dose 4
Description: as for outcome 5
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51776 | 5164
Events per 1000 person-days | 0.019 [0.003 to 0.137] | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

51. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 7 Days After Dose 4
Description: as for outcome 6
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 103551 | 10328
Events per 1000 person-days | 0.010 [0.001 to 0.069] | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

52. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 3 Days After Dose 4
Description: as for outcome 7
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51741 | 5160
Events per 1000 person-days
  Urticaria | 0.29 [0.175 to 0.481] | 0.388 [0.097 to 1.550]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

53. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 4 to 7 Days After Dose 4
Description: as for outcome 8
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51727 | 5164
Events per 1000 person-days
  Urticaria | 0.483 [0.327 to 0.715] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

54. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 7 Days After Dose 4
Description: as for outcome 9
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 103407 | 10316
Events per 1000 person-days
  Urticaria | 0.387 [0.284 to 0.527] | 0.194 [0.049 to 0.775]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

55. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 3 Days After Dose 4
Description: as for outcome 10
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51776 | 5164
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

56. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 4 to 7 Days After Dose 4
Description: as for outcome 12
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51776 | 5164
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

57. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 7 Days After Dose 4
Description: as for outcome 12
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 103552 | 10328
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

58. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 3 Days After Dose 4
Description: as for outcome 13
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51641 | 4930
Events per 1000 person-days | 1.278 [1.004 to 1.627] | 15.822 [12.673 to 19.753]

59. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 4 to 7 Days After Dose 4
Description: as for outcome 14
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 51622 | 5121
Events per 1000 person-days | 1.298 [1.022 to 1.649] | 3.124 [1.914 to 5.1]

60. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 7 Days After Dose 4
Description: as for outcome 15
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Person days at risk) | 103028 | 9749
Events per 1000 person-days | 1.194 [1.001 to 1.425] | 9.54 [7.785 to 11.690]

61. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 3 Days After All Doses
Description: as for outcome 1
Time Frame: 0 to 3 Days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284246 | 31364
Events per 1000 person-days | 0.011 [0.003 to 0.033] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

62. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 4 to 7 Days After All Doses
Description: as for outcome 2
Time Frame: 4 to 7 Days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284252 | 31364
Events per 1000 person-days | 0.014 [0.005 to 0.038] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

63. Primary Outcome: Incidence Rate (Per 1000 Person Days) of All Seizures Through 0 to 7 Days After All Doses
Description: as for outcome 3
Time Frame: 0 to 7 Days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 568486 | 62728
Events per 1000 person-days | 0.012 [0.006 to 0.026] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

64. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 3 Days After All Doses
Description: as for outcome 4
Time Frame: 0 to 3 Days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284256 | 31364
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had febrile seizures during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizures during the specified risk window.

65. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 4 to 7 Days After All Doses
Description: as for outcome 5
Time Frame: 4 to 7 Days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284254 | 31364
Events per 1000 person-days | 0.007 [0.002 to 0.028] | NA [NA to NA] — Data was not estimable as no participant had febrile seizures during the specified risk window.

66. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Febrile Seizures Through 0 to 7 Days After All Doses
Description: as for outcome 6
Time Frame: 0 to 7 Days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 568510 | 62728
Events per 1000 person-days | 0.004 [0.001 to 0.014] | NA [NA to NA] — Data was not estimable as no participant had febrile seizures during the specified risk window.

67. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 3 Days After All Doses
Description: as for outcome 7
Time Frame: 0 to 3 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284202 | 31353
Events per 1000 person-days
  Urticaria | 0.088 [0.059 to 0.130] | 0.223 [0.106 to 0.468]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

68. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 4 to 7 Days After All Doses
Description: as for outcome 8
Time Frame: 4 to 7 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284162 | 31364
Events per 1000 person-days
  Urticaria | 0.165 [0.124 to 0.220] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

69. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Urticaria and Angioedema Through 0 to 7 Days After All Doses
Description: as for outcome 9
Time Frame: 0 to 7 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 568263 | 62689
Events per 1000 person-days
  Urticaria | 0.127 [0.101 to 0.160] | 0.112 [0.053 to 0.234]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

70. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 3 Days After All Doses
Description: as for outcome 10
Time Frame: 0 to 3 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284256 | 31364
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

71. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 4 to 7 Days After All Doses
Description: as for outcome 11
Time Frame: 4 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284256 | 31364
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

72. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Apnea Through 0 to 7 Days After All Doses
Description: as for outcome 12
Time Frame: 0 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 568512 | 62728
Events per 1000 person-days | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

73. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 3 Days After All Doses
Description: as for outcome 13
Time Frame: 0 to 3 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 283817 | 30628
Events per 1000 person-days | 0.627 [0.542 to 0.726] | 7.575 [6.660 to 8.615]

74. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 4 to 7 Days After All Doses
Description: as for outcome 14
Time Frame: 4 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 284051 | 31303
Events per 1000 person-days | 0.331 [0.270 to 0.405] | 0.958 [0.67 to 1.371]

75. Primary Outcome: Incidence Rate (Per 1000 Person Days) of Fever Through 0 to 7 Days After All Doses
Description: as for outcome 15
Time Frame: 0 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Units Other Than Participants: Person days at risk
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Person days at risk) | 567188 | 61016
Events per 1000 person-days | 0.458 [0.406 to 0.518] | 4.261 [3.774 to 4.812]

76. Primary Outcome: Incidence Rate (IR) (Per 1000 Doses) of All Seizures Through 0 to 3 Days After Dose 1
Description: IR was calculated as the number of all seizure events experienced during the specified risk window (0-3 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

77. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of all seizure events experienced during the specified risk window (4-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | 0.098 [0.025 to 0.394] | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

78. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of all seizure events experienced during the specified risk window (0-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | 0.098 [0.025 to 0.394] | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

79. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of febrile seizure events experienced during the specified risk window (0-3 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

80. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of febrile seizure events experienced during the specified risk window (4-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | 0.049 [0.007 to 0.349] | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

81. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of febrile seizure events experienced during the specified risk window (0-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | 0.049 [0.007 to 0.349] | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

82. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of urticaria and angioedema events experienced during the specified risk window (0-3 days post-vaccination) divided by the number of doses, multiply by 1000. Urticaria represents an allergic reaction. Angioedema is an area of swelling (edema) of the lower layer of skin and tissue just under the skin or mucous membranes.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses
  Urticaria | 0.049 [0.007 to 0.349] | 1.304 [0.421 to 4.044]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

83. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of urticaria and angioedema events experienced during the specified risk window (4-7 days post-vaccination) divided by the number of doses, multiply by 1000. Urticaria represents an allergic reaction. Angioedema is an area of swelling (edema) of the lower layer of skin and tissue just under the skin or mucous membranes.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses
  Urticaria | 0.098 [0.025 to 0.394] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

84. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of urticaria and angioedema events experienced during the specified risk window (0-7 days post-vaccination) divided by the number of doses, multiply by 1000. Urticaria represents an allergic reaction. Angioedema is an area of swelling (edema) of the lower layer of skin and tissue just under the skin or mucous membranes.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses
  Urticaria | 0.148 [0.048 to 0.458] | 1.304 [0.421 to 4.044]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

85. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of apnea events experienced during the specified risk window (0-3 days post-vaccination) divided by the number of doses, multiply by 1000. Apnea is the cessation of breathing.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

86. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of apnea events experienced during the specified risk window (4-7 days post-vaccination) divided by the number of doses, multiply by 1000. Apnea is the cessation of breathing.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

87. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of apnea events experienced during the specified risk window (0-7 days post-vaccination) divided by the number of doses, multiply by 1000. Apnea is the cessation of breathing.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

88. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 3 Days After Dose 1
Description: Incidence rate was calculated as the number of fever events experienced during the specified risk window (0-3 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 3 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | 2.215 [1.654 to 2.966] | 41.304 [33.780 to 50.504]

89. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 4 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of fever events experienced during the specified risk window (4-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 4 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | 0.197 [0.074 to 0.525] | 2.174 [0.905 to 5.223]

90. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 7 Days After Dose 1
Description: Incidence rate was calculated as the number of fever events experienced during the specified risk window (0-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 7 days after Dose 1
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 20318 | 2300
Events per 1000 doses | 2.362 [1.780 to 3.135] | 43.478 [35.74 to 52.892]

91. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 3 Days After Dose 2
Description: Incidence rate was calculated as the number of all seizure events experienced during the specified risk window (0-3 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

92. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 4 to 7 Days After Dose 2
Description: as for outcome 77
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

93. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 7 Days After Dose 2
Description: as for outcome 78
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

94. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 3 Days After Dose 2
Description: as for outcome 79
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

95. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 4 to 7 Days After Dose 2
Description: as for outcome 80
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

96. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 7 Days After Dose 2
Description: as for outcome 81
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

97. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 3 Days After Dose 2
Description: as for outcome 82
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses
  Urticaria | 0.258 [0.107 to 0.620] | 0.908 [0.227 to 3.630]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

98. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 4 to 7 Days After Dose 2
Description: as for outcome 83
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses
  Urticaria | 0.516 [0.278 to 0.959] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

99. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 7 Days After Dose 2
Description: as for outcome 84
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses
  Urticaria | 0.774 [0.466 to 1.283] | 0.908 [0.227 to 3.630]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

100. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 3 Days After Dose 2
Description: as for outcome 85
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

101. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 4 to 7 Days After Dose 2
Description: as for outcome 86
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

102. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 7 Days After Dose 2
Description: as for outcome 87
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

103. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 3 Days After Dose 2
Description: as for outcome 88
Time Frame: 0 to 3 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | 2.063 [1.513 to 2.813] | 16.341 [11.788 to 22.655]

104. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 4 to 7 Days After Dose 2
Description: as for outcome 89
Time Frame: 4 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | 0.464 [0.242 to 0.892] | 2.270 [0.945 to 5.453]

105. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 7 Days After Dose 2
Description: as for outcome 90
Time Frame: 0 to 7 days after Dose 2
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 19387 | 2203
Number analyzed (Doses) | 19387 | 2203
Events per 1000 doses | 2.476 [1.866 to 3.285] | 18.611 [13.704 to 25.276]

106. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 3 Days After Dose 3
Description: as for outcome 91
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

107. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 4 to 7 Days After Dose 3
Description: as for outcome 77
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

108. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 7 Days After Dose 3
Description: as for outcome 78
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had seizure during the specified risk window.

109. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 3 Days After Dose 3
Description: as for outcome 79
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

110. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 4 to 7 Days After Dose 3
Description: as for outcome 80
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

111. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 7 Days After Dose 3
Description: as for outcome 81
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

112. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 3 Days After Dose 3
Description: as for outcome 82
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses
  Urticaria | 0.217 [0.082 to 0.579] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

113. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 4 to 7 Days After Dose 3
Description: as for outcome 83
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses
  Urticaria | 0.543 [0.292 to 1.009] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

114. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 7 Days After Dose 3
Description: as for outcome 84
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses
  Urticaria | 0.760 [0.450 to 1.284] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

115. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 3 Days After Dose 3
Description: as for outcome 85
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

116. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 4 to 7 Days After Dose 3
Description: as for outcome 86
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

117. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 7 Days After Dose 3
Description: as for outcome 87
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

118. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 3 Days After Dose 3
Description: as for outcome 88
Time Frame: 0 to 3 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | 1.466 [1.006 to 2.138] | 11.236 [7.467 to 16.908]

119. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 4 to 7 Days After Dose 3
Description: as for outcome 89
Time Frame: 4 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | 0.760 [0.450 to 1.284] | 1.954 [0.733 to 5.207]

120. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 7 Days After Dose 3
Description: as for outcome 90
Time Frame: 0 to 7 days after Dose 3
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 18415 | 2047
Number analyzed (Doses) | 18415 | 2047
Events per 1000 doses | 2.226 [1.639 to 3.024] | 12.702 [8.648 to 18.655]

121. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 3 Days After Dose 4
Description: as for outcome 91
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | 0.232 [0.075 to 0.719] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

122. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 4 to 7 Days After Dose 4
Description: Incidence rate was calculated as the number of all seizures events experienced during the specified risk window (4-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | 0.155 [0.039 to 0.618] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

123. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 7 Days After Dose 4
Description: Incidence rate was calculated as the number of all seizures events experienced during the specified risk window (0-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | 0.386 [0.161 to 0.928] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

124. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 3 Days After Dose 4
Description: as for outcome 79
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

125. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 4 to 7 Days After Dose 4
Description: as for outcome 80
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | 0.077 [0.011 to 0.548] | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

126. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 7 Days After Dose 4
Description: as for outcome 81
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | 0.077 [0.011 to 0.548] | NA [NA to NA] — Data was not estimable as no participant had febrile seizure during the specified risk window.

127. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 3 Days After Dose 4
Description: as for outcome 82
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses
  Urticaria | 1.159 [0.699 to 1.922] | 1.549 [0.387 to 6.194]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

128. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 4 to 7 Days After Dose 4
Description: as for outcome 83
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses
  Urticaria | 1.931 [1.305 to 2.858] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

129. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 7 Days After Dose 4
Description: as for outcome 84
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses
  Urticaria | 3.090 [2.267 to 4.213] | 1.549 [0.387 to 6.194]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

130. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 3 Days After Dose 4
Description: as for outcome 85
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

131. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 4 to 7 Days After Dose 4
Description: as for outcome 86
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

132. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 7 Days After Dose 4
Description: as for outcome 87
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

133. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 3 Days After Dose 4
Description: as for outcome 88
Time Frame: 0 to 3 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | 5.099 [4.006 to 6.490] | 60.418 [48.394 to 75.431]

134. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 4 to 7 Days After Dose 4
Description: as for outcome 89
Time Frame: 4 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | 5.176 [4.074 to 6.577] | 12.394 [7.593 to 20.230]

135. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 7 Days After Dose 4
Description: as for outcome 90
Time Frame: 0 to 7 days after Dose 4
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 12944 | 1291
Number analyzed (Doses) | 12944 | 1291
Events per 1000 doses | 9.503 [7.963 to 11.339] | 72.037 [58.788 to 88.272]

136. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 3 Days After All Doses
Description: Incidence rate was calculated as the number of all seizures events experienced during the specified risk window (0-3 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 3 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | 0.042 [0.014 to 0.131] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

137. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 4 to 7 Days After All Doses
Description: as for outcome 122
Time Frame: 4 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | 0.056 [0.021 to 0.15] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

138. Primary Outcome: Incidence Rate (Per 1000 Doses) of All Seizures Through 0 to 7 Days After All Doses
Description: as for outcome 123
Time Frame: 0 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | 0.099 [0.047 to 0.207] | NA [NA to NA] — Data was not estimable as no participant had seizures during the specified risk window.

139. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 3 Days After All Doses
Description: Incidence rate was calculated as the number of febrile seizures events experienced during the specified risk window (0-3 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 3 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had febrile seizures during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had febrile seizures during the specified risk window.

140. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 4 to 7 Days After All Doses
Description: Incidence rate was calculated as the number of febrile seizures events experienced during the specified risk window (4-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 4 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | 0.028 [0.007 to 0.113] | NA [NA to NA] — Data was not estimable as no participant had febrile seizures during the specified risk window.

141. Primary Outcome: Incidence Rate (Per 1000 Doses) of Febrile Seizures Through 0 to 7 Days After All Doses
Description: Incidence rate was calculated as the number of febrile seizures events experienced during the specified risk window (0-7 days post-vaccination) divided by the number of doses, multiply by 1000.
Time Frame: 0 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | 0.028 [0.007 to 0.113] | NA [NA to NA] — Data was not estimable as no participant had febrile seizures during the specified risk window.

142. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 3 Days After All Doses
Description: as for outcome 82
Time Frame: 0 to 3 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses
  Urticaria | 0.352 [0.238 to 0.521] | 0.893 [0.426 to 1.873]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

143. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 4 to 7 Days After All Doses
Description: as for outcome 83
Time Frame: 4 to 7 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses
  Urticaria | 0.661 [0.497 to 0.880] | NA [NA to NA] — Data was not estimable as no participant had urticaria during the specified risk window.
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

144. Primary Outcome: Incidence Rate (Per 1000 Doses) of Urticaria and Angioedema Through 0 to 7 Days After All Doses
Description: as for outcome 84
Time Frame: 0 to 7 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses
  Urticaria | 1.013 [0.804 to 1.276] | 0.893 [0.426 to 1.873]
  Angioedema | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had angioedema during the specified risk window.

145. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 3 Days After All Doses
Description: as for outcome 85
Time Frame: 0 to 3 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

146. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 4 to 7 Days After All Doses
Description: as for outcome 86
Time Frame: 4 to 7 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

147. Primary Outcome: Incidence Rate (Per 1000 Doses) of Apnea Through 0 to 7 Days After All Doses
Description: as for outcome 87
Time Frame: 0 to 7 days after all Doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window. | NA [NA to NA] — Data was not estimable as no participant had apnea during the specified risk window.

148. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 3 Days After All Doses
Description: as for outcome 88
Time Frame: 0 to 3 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | 2.505 [2.163 to 2.901] | 29.588 [26.016 to 33.651]

149. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 4 to 7 Days After All Doses
Description: as for outcome 89
Time Frame: 4 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | 1.323 [1.081 to 1.619] | 3.826 [2.675 to 5.472]

150. Primary Outcome: Incidence Rate (Per 1000 Doses) of Fever Through 0 to 7 Days After All Doses
Description: as for outcome 90
Time Frame: 0 to 7 days after all doses
Population: Analysis population included all participants included in the main study cohort and prospective cohort respectively.
Measure: Number (95% Confidence Interval); unit: Events per 1000 doses
Units Other Than Participants: Doses
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
Number analyzed (Participants) | 20318 | 2300
Number analyzed (Doses) | 71064 | 7841
Events per 1000 doses | 3.659 [3.240 to 4.132] | 33.159 [29.364 to 37.445]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to the nature of claims database from which data were queried, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not meet, hence adverse events were not collected and reported.
Arm/Group | Prevenar 13: Main Study Cohort | Prevenar 13 Cohort: Prospective Cohort Study
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT03656939/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT03656939/SAP_001.pdf